CLINICAL TRIAL: NCT01805830
Title: Phase III, Double Blind, Parallel-group, Randomized, Placebo Controlled Study to Compare the Efficacy and Safety of MP-513 When Added to Ongoing Metformin Monotherapy In Patients With Type 2 DM
Brief Title: Teneligliptin(MP-513) vs. Placebo in Patient With Metformin Monotherapy
Acronym: T2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP_C301
Record Dates: First submitted 2012-12-26; First posted 2013-03-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes
Keywords: Type2DM / DPP-IV inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MP513 group (Experimental)
  Interventions: Drug: MP513
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP513 — form : Pink film-coated tablet for oral administration Dosage : 20mg/tablet frequency and duration: 1 tablet/day
  Arms: MP513 group
Drug: Placebo — form : Pink film-coated tablet for oral administration Dosage : 20mg/tablet frequency and duration: 1 tablet/day
  Arms: Placebo group

SUMMARY:
The study design of this trial is double blind, parallel-group, randomized, Placebo controlled study.

DETAILED DESCRIPTION:
* Although many different oral antidiabetic agents are currently available, approximately 50% of treated Type 2 diabetic subjects do not reach currently accepted goals for HbA1c(Oral communication, American Diabetic Association, 2008)
* Subjects are frequently prescribed agents which can cause hypoglycemia, and/or weight gain. Metformin does not usually have these unwanted effects, and it is the standard first line therapy in treating type 2 diabetic mellitus in European union.
* Nonclinical pharmacodynamic studies revealed that MP-513 effectively improves glucose tolerance in animal models of type 2 diabetes, whilst the compound has very little potential to cause hypoglycaemia, the most commonly reported adverse event with many currently marketed products.
* The nonclinical studies also suggested that the inhibitory effect of MP-513 on DPP-Ⅳ is more potent and durable than other DPP-Ⅳ inhibitors in development. The result in safety pharmacology and toxicology also revealed that MP-513 has a relatively wide margin for safety.
* Thus, MP-513 is expected to have good efficacy and tolerability in subjects with type 2 diabetes mellitus by once-daily administration.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged ≥18 years at signature of the ICF
2. The subject has had a documented diagnosis of Type 2 diabetes for at least 6 months at the screening visit
3. The subject's Type 2 diabetes is managed by metformin monotherapy ≥1000 mg/day, plus diet and exercise, as appropriate, and the dose has been unchanged for at least 56 consecutive days
4. The subject's HbA1c is 7.0%≤HbA1c<10.0%
5. The subject's BMI is 20.0≤BMI≤40.0kg/m2
6. The subject's FPG is <15 mmol/L (270 mg/dL)
7. The subject is capable of giving informed consent, complying with the restrictions and requirements of the protocol

Exclusion Criteria:

1. The subject is suffering from any disease, including Type 2 diabetes or its complications that, in the opinion of the Investigator, is sufficiently severe to render the subject unfit, or affect the subject's ability, to participate in the study, for example:

   * Macroangiopathy with symptoms of coronary heart disease or peripheral arterial obstructive disease.
   * Microangiopathy with symptoms of (autonomous) neuropathy with any one or more of the following: gastroparesis
   * Symptoms of poor blood glucose control (polyuria, polydipsia or weight loss)
2. The subject has a history of Type 1 diabetes or a secondary form of diabetes
3. The subject has a history of allergy to MP-513, or to any of the excipients in the MP-513 tablet (eg. Mannitol)
4. The subject has a history of drug abuse
5. The subject drinks on average more than 28 units of alcohol per week(One unit of alcohol equals approximately 250 mL of beer, 125 mL of wine or 40 mL of spirits)
6. The subject has a medical history of unstable angina, or heart failure(New York Heart Association class Ⅲ-IV) or any clinically significant ECG abnormalities such as ventricular tachycardia or a medical history of ventricular tachycardia
7. The subject has participated in any other clinical study involving blood draws or administration of an unlicensed medicinal product within 12 weeks prior to the screening visit (This does not preclude a subject from being re-screened for this study at a later date within the 12 week period, provided they were not randomised )
8. The subject has received insulin within 12 months prior to the screening visit, with the exception of insulin therapy during hospitalization, insulin therapy for medical conditions not requiring hospitalization (<2 weeks duration) or use in gestational diabetes
9. The subject is suffering from serious concurrent renal disease or creatinine clearance <60 mL/min
10. Non-surgically sterilised, pre-menopausal female subject, who does not agree to use a double barrier method of contraception from the screening visit until at least 14 days after the last dosing day (Examples of permitted types of contraception are: condoms, cervical cap in conjunction with spermicide, sterilisation and intra-uterine device. Oral contraception is permitted but must not be used as the sole method of contraception)
11. Female subjects whose pregnancy test is negative or who are pregnant, lactating, or are planning to become pregnant during the study
12. The subject is expected to require additional diabetic treatment for his/her Type 2 diabetes or its complications during the study after the screening visit
13. The subject has a clinically significant liver disease with aspartate-amino-transferase (AST) and alanine-amino-transferase (ALT) >2.5 times the upper limit of normal (ULN) at the screening visit
14. The subject has diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg at the screening visit
15. The presence of any other condition that leads the investigator to conclude that the patient is inappropriate for inclusion in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from Visit 1(Baseline Visit) in HbA1c at Visit 5(week 16)

SECONDARY OUTCOMES:
FPG(Fasting Plasma Glucose) | Change from Visit 1(Baseline Visit) in FPG at Visit 5(week 16)
Weight | Change from Visit 1(Baseline Visit) in weight at Visit 5(week 16)
BMI | Change from Visit 1(Baseline Visit) in BMI at Visit 5(week 16)
HbA1c <7.0% | The proportion of patients who achieve an HbA1c<7.0% at Visit 5(week 16)
HbA1c <6.5% | The proportion of patients who achieve an HbA1c<6.5% at Visit 5(week 16)
Total Cholesterol | Change from Visit 1(Baseline Visit) in Total Cholesterol at Visit 5(week 16)
LDL Cholesterol | Change from Visit 1(Baseline Visit) in LDL Cholesterol at Visit 5(week 16)
HDL Cholesterol | Change from Visit 1(Baseline Visit) in HDL Cholesterol at Visit 5(week 16)
Triglyceride | Change from Visit 1(Baseline Visit) in Triglyceride at Visit 5(week 16)
C-peptide | Change from Visit 1(Baseline Visit) in C-peptide at Visit 5(week 16)
Insulin | Change from Visit 1(Baseline Visit) in insulin at Visit 5(week 16)
hsCRP | Change from Visit 1(Baseline Visit) in hsCRP at Visit 5(week 16)
HOMA-β | Change from Visit 1(Baseline Visit) in HOMA-β at Visit 5(week 16)
HOMA-IR | Change from Visit 1(Baseline Visit) in HOMA-IR at Visit 5(week 16)

CONTACTS AND LOCATIONS:
Overall Officials: BONGYUN CHA, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Handok Pharmaceuticals CO. LTD, Seoul, Seoul, South Korea